CLINICAL TRIAL: NCT07361068
Title: Evaluation of Intraoperative Cerebral Desaturation and Risk Factors Associated With Cognitive Dysfunction After Cardiac Surgery
Brief Title: Assessment of Brain Oxygen Drops During Surgery and Related Risk Factors for Cognitive Problems After Heart Surgery
Status: Completed | Type: Observational
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, ŞULE BALK, Anesthesiology and Reanimation doctor, Bursa Yuksek Ihtisas Training and Research Hospital
Other Study IDs: 011-KAEK-25 2023/02-15
Record Dates: First submitted 2025-12-22; First posted 2026-01-22 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Cognitive Dysfunction, Postoperative; Cognitive Dysfunction; Cardiac Surgery
Keywords: Cognitive dysfunction; Near infrared spectroscopy; cardiopulmonary bypass
MeSH Terms: conditions — Postoperative Cognitive Complications; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group POCD: Patients develop cognitive dysfunction after cardiac surgery: The POCD group (n=24) comprised patients undergoing elective cardiac surgery with cardiopulmonary bypass who developed postoperative cognitive dysfunction, defined as an MMSE score ≤23 at any postoperative assessment. ( Postoperative day 4 ,7, 30)
- Group non-POCD : Patients did not develop postoperative cognitive dysfunction: The non-POCD group (n = 50) consisted of adult patients undergoing elective cardiac surgery with cardiopulmonary bypass whose MMSE scores remained ≥24 at all postoperative assessments, indicating no postoperative cognitive dysfunction.

SUMMARY:
This study examines whether decreases in brain oxygen levels during cardiac surgery are linked to postoperative cognitive dysfunction and identifies other factors that may increase the risk of cognitive impairment.

DETAILED DESCRIPTION:
In this prospective study, the relationship between intraoperative cerebral oxygen saturation and postoperative cognitive dysfunction (POCD) was investigated in adult patients undergoing elective cardiac surgery with cardiopulmonary bypass (CPB). Patients with a preoperative Mini-Mental State Examination (MMSE) score ≥ 24, no history of cerebrovascular disease, and no conditions that could interfere with near-infrared spectroscopy (NIRS) monitoring were included.

Measurements were recorded at the following time points: T0 (before induction), T1 (15 minutes after induction), T2 (5 minutes after initiation of CPB), T3 (during the hypothermic phase of CPB), T4 (rewarming phase of CPB, at 34 °C), T5 (termination of CPB), and T6 (upon admission to the intensive care unit). Patients were divided into two groups according to postoperative cognitive outcomes: those who developed POCD and those who did not.

Cognitive function was assessed using the MMSE preoperatively and on postoperative days 4, 7, and 30. During surgery, cerebral oxygen saturation was measured at predefined time points using NIRS probes placed on the frontal region, and detailed intraoperative and perioperative data were recorded. Standardized interventions were implemented when a decrease of more than 20% in regional cerebral oxygen saturation (rSO₂) from baseline was detected in order to maintain adequate cerebral oxygenation.

ELIGIBILITY:
Inclusion Criteria:

* Planned elective CPB surgery
* Provision of written informed consent
* Absence of communication barriers that could interfere with preoperative and postoperative MMSE assessment
* No history of cerebrovascular disease
* Preoperative MMSE score ≥24
* Education level of at least high school
* Absence of any frontal deformity that could hinder NIRS monitoring

Exclusion Criteria:

* Preoperative use of antipsychotic or antidepressant medications
* Emergency cardiac surgery indication
* Presence of ≥50% carotid artery stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing open heart surgery with cardiopulmonary bypass under general anesthesia
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
Incidence of Postoperative Cognitive Dysfunction (POCD) | Baseline (preoperative, before surgery) and postoperative day 4, postoperative day 7, and postoperative day 30.
  Postoperative cognitive dysfunction (POCD) is defined as a decline in cognitive performance assessed using the Mini-Mental State Examination (MMSE), with a score of ≤23 at any postoperative assessment compared with a preoperative baseline MMSE score of ≥24. This primary outcome evaluates the association between intraoperative cerebral oxygen desaturation, measured by near-infrared spectroscopy (NIRS) as a reduction of >20% from baseline regional cerebral oxygen saturation (rSO₂), and postoperative cognitive dysfunction following cardiac surgery with cardiopulmonary bypass.

SECONDARY OUTCOMES:
Intraoperative Cerebral Oxygen Desaturation Measured by NIRS | Perioperatively (during surgery) through immediate postoperative period (upon ICU admission).
  Magnitude of intraoperative decreases in regional cerebral oxygen saturation (rSO₂) relative to baseline, measured using near-infrared spectroscopy (NIRS) at predefined intraoperative time points.
  Measurements are recorded at:
  T0: before induction of anesthesia T1: 15 minutes after induction of anesthesia T2: 5 minutes after initiation of cardiopulmonary bypass (CPB) T3: hypothermic phase of CPB T4: rewarming phase of CPB (34 °C) T5: weaning from CPB T6: upon admission to the intensive care unit (ICU)
Postoperative Cognitive Performance Over Time Assessed by MMSE | Baseline (preoperative, before surgery) and postoperative day 4, postoperative day 7, and postoperative day 30.
  Changes in cognitive performance over time assessed using the Mini-Mental State Examination (MMSE) to evaluate early and late postoperative cognitive recovery.
Operation Time | From skin incision to skin closure during surgery
  Operation time will be compared between patients with and without postoperative cognitive dysfunction (POCD).
  Measure : Minute
Cardiopulmonary Bypass (CPB) Duration | From initiation to termination of cardiopulmonary bypass during surgery (single intraoperative assessment).
  Cardiopulmonary bypass duration will be compared between patients with and without postoperative cognitive dysfunction (POCD).
  Measure : Minute
Aortic Cross-Clamp (ACC) Duration | From application to removal of the aortic cross-clamp during surgery (single intraoperative assessment)
  Aortic cross-clamp duration will be compared between patients with and without postoperative cognitive dysfunction (POCD).
  Meusure: Minute
Time to Extubation | From completion of surgery until successful extubation, assessed up to 30 postoperative days
  Time to extubation will be compared between patients with and without postoperative cognitive dysfunction (POCD).
  Measure: Hour
Intensive Care Unit Length of Stay | From ICU admission after surgery until ICU discharge, assessed up to 30 postoperative days.
  Length of intensive care unit stay will be compared between patients with and without postoperative cognitive dysfunction (POCD).
  Measure: Hour
Hospital Length of Stay | From hospital admission for cardiac surgery until hospital discharge, assessed up to 30 postoperative days.
  Hospital length of stay will be compared between patients with and without postoperative cognitive dysfunction (POCD).
  Measure: Day
Correlation Between Perioperative Clinical Variables and Postoperative MMSE Scores | Postoperative day 4, postoperative day 7, and postoperative day 30.
  Correlation between perioperative clinical variables and postoperative cognitive performance assessed using the Mini-Mental State Examination (MMSE). Variables correlated with MMSE scores include: Operation time (minutes) Cardiopulmonary bypass (CPB) duration (minutes) Aortic cross-clamp (ACC) duration (minutes) Intensive care unit (ICU) length of stay (hours) Hospital length of stay (days)

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Yuksek Ihtisas Traning and Research Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Hu YN, Hsieh TH, Tsai MT, Chien CY, Roan JN, Huang YC, Liang SF. Cognitive Function Deterioration After Cardiopulmonary Bypass: Can Intraoperative Optimal Cerebral Regional Tissue Oxygen Saturation Predict Postoperative Cognitive Function? J Cardiothorac Vasc Anesth. 2023 May;37(5):715-723. doi: 10.1053/j.jvca.2023.01.025. Epub 2023 Feb 2. PMID 36813631
- [Result] Lewis C, Parulkar SD, Bebawy J, Sherwani S, Hogue CW. Cerebral Neuromonitoring During Cardiac Surgery: A Critical Appraisal With an Emphasis on Near-Infrared Spectroscopy. J Cardiothorac Vasc Anesth. 2018 Oct;32(5):2313-2322. doi: 10.1053/j.jvca.2018.03.032. Epub 2018 Mar 20. PMID 30100271